CLINICAL TRIAL: NCT05997225
Title: Preventing Lung Cancer Through Tobacco Cessation at FDNY
Brief Title: Tobacco Cessation at FDNY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: FDNY World Trade Center Health Program (Unknown); National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-14980; R21OH012256 (NIH)
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Tobacco Use; Tobacco Smoking; Tobacco Use Cessation
Keywords: World Trade Center Health Program; occupational medicine; tobacco cessation; lifestyle medicine; opt-out treatment
MeSH Terms: conditions — Tobacco Use; Tobacco Smoking; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enhanced Care (Experimental): Opt-out counseling enrollment. individually-tailored biofeedback linked to Chest CT and spirometry results.
  Varenicline: Preloading regimen (prior to target quit date): 0.5 mg once a day for days 1-3, 0.5 mg twice a day for days 4-7, and 1 mg twice a day for days 8-28.
  1 mg twice day for 12 weeks after target quit date.
  Interventions: Other: opt out enrollment, tailored counseling, varenicline started prior to target quit date
- Standard Care (Active Comparator): Opt-in counseling enrollment. Standard tobacco cessation counseling.
  Varenicline: Preloading regimen (prior to target quit date): 0.5 mg once a day for days 1-3, 0.5 mg twice a day for days 4-7, and 1 mg twice a day for days 8-28.
  1 mg twice day for 12 weeks after target quit date.
  Interventions: Other: opt in enrollment, non-tailored counseling, varenicline started prior to target quit date

INTERVENTIONS:
Other: opt out enrollment, tailored counseling, varenicline started prior to target quit date — Participants automatically enrolled in motivational counseling. Tailored counseling includes sharing results of Chest CT results and lung function spirometry tests with participants.
  Arms: Enhanced Care
Other: opt in enrollment, non-tailored counseling, varenicline started prior to target quit date — Participants must opt-in to receive counseling. Counseling does not include discussion of Chest CT or spirometry results.
  Arms: Standard Care

SUMMARY:
At the Fire Department of the City of New York (FDNY) World Trade Center Health Program, 36% of participants in the low dose computed tomography (LDCT) lung cancer screening program are current smokers, despite referral to the free FDNY Tobacco Cessation Program (Standard Care). Investigators propose testing an Enhanced Care program which includes opt-out enrollment; tobacco cessation counseling will be individually tailored to spirometry/LDCT results and treatment with varenicline starting 4 weeks prior to their target quit date. This randomized trial will compare enrollment and cessation outcomes in Standard Care vs. Enhanced Care groups of challenging-to-treat, high-risk smokers.

DETAILED DESCRIPTION:
The overarching goal of this Randomized Controlled trial is to develop and test an effective, scalable intervention with potential to reach high-risk smokers undergoing CT lung cancer screening who have not engaged in or succeeded with traditional tobacco treatment approaches. The investigators will test an Enhanced Care intervention specifically designed to address multiple challenges to tobacco treatment engagement and success. First, the researchers will test opt-out enrollment in cessation treatment. The current tobacco treatment default, in which patients must opt-in to cessation treatment and are only offered counseling and pharmacotherapy when deemed ready to quit, results in missed opportunities to engage smokers into treatment. Previous studies of opt-out enrollment in cessation treatment suggest that an opt-out tobacco treatment strategy substantially increases engagement and cessation rates compared with traditional opt-in approaches. Second, proactive counseling will leverage the "reachable, teachable moment" of CT screening to motivate cessation through individually tailored messaging tied to CT results and lung function spirometry. Using CT results as a motivational tool has shown promise in pilot studies. The optimal approach and success of using CT coupled with spirometry results to motivate tobacco cessation remains unknown. Third, investigators will offer varenicline pre-loading to all enrollees, regardless of study arm, in which varenicline is initiated 4 weeks prior to target quit date. This approach is associated with decreased pre-quit tobacco-associated reward and double the rate of abstinence compared with standard varenicline treatment.

The investigators thus propose a randomized trial among retired FDNY World Trade Center Health Program responders eligible for the FDNY World Trade Center Health Program CT screening program to test the effects of Enhanced Care (opt-out enrollment, tailored counseling based on CT and spirometry results, and varenicline with preloading) against Standard Care (opt-in enrollment, standard cessation counseling without spirometry/CT tailoring, and varenicline with preloading) in the engagement of high-risk smokers in cessation treatment and the achievement of tobacco abstinence.

ELIGIBILITY:
Inclusion Criteria

* Enrolled in FDNY World Trade Center Health Program (WTCHP)
* Retired
* Age ≥ 50 years old
* Self-reported current smoker on most recent questionnaire OR self-reported current smoker in the past 5 years
* 20 pack-year smoker OR 20-year smoking duration

Exclusion Criteria

* Reduced renal function
* estimated glomerular filtration rate (eGFR) <30 [CKD-EPI Creatinine Equation (2021)] at last World Trade Center (WTC) medical monitoring blood exam OR ICD10 codes for kidney disease: N04.9, N17.9, N18.9, Z94.0, E13.21, N18.9, I12.9, N00.9, N03.9
* Undergoing active cancer treatment, defined as being diagnosed on 1/1/2022 or later
* Clinical instability (e.g., hospitalization in last 3 months)
* Using varenicline in last 30 days
* Endorsing suicidal ideations: moderate or high risk on Columbia-Suicide Severity Rating Scale (C-SSRS)
* Screened for alcohol use disorder AUDIT>15

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Enrollment | Baseline (Week 0)
  Enrollment is defined as first visit attendance with our tobacco treatment specialist in FDNY's Tobacco Cessation Program: Standard vs. Enhanced Care arms. The number of participants who attend the first visit with the tobacco treatment specialist will be tabulated and reported.
Tobacco Abstinence | From baseline (Week 0) through each research assessment visit up to the 12-week post EOT timepoint visit at 28 weeks
  7-day point prevalence abstinence will be biochemically verified by the analysis of urine samples collected at a laboratory nearest each participant's residence. Urine samples collection will occur at baseline, and at weeks 2, 4, 8, 12, and 16 along with a 12-week post end of treatment (EOT) timepoint at 28 weeks. Samples will be analyzed for urine cotinine which is the commonly measured biomarker of nicotine intake. Urine cotinine levels < 20 ng/mL will be used to verify tobacco abstinence. Data will be summarized at each timepoint by study arm using basic descriptive statistics at each research assessment visit.

SECONDARY OUTCOMES:
Retention to Study End-Date | Through the 12-week post EOT timepoint at 28 weeks
  Retention will be assessed and reported as the number of participants retained in the study through the time of the 12-week post end of treatment (EOT) timepoint at 28 weeks.
Counseling adherence | From baseline (Week 0) through each visit up to the 12-week post EOT timepoint visit at 28 weeks
  Counseling adherence will be determined by the number of counseling visits attended. Tobacco counseling sessions will occur at baseline, and at weeks 2, 4, 8, 12, and 16 along with a 12-week post end of treatment (EOT) timepoint at 28 weeks. Counseling adherence will be summarized by study arm based on attendance during each individual session (timepoint) and reported as a continuous variable for each timepoint (counseling visit).
Varenicline (pill count) adherence | Up through the time of the final research visit at Week 16
  Varenicline adherence will be measured using pill counts, recorded as the pills taken / pills prescribed (i.e., the number of pills taken divided by the number of pills prescribed) per participant, corresponding to the dosing regimen. Varenicline adherence data will be summarized by study arm using basic descriptive statistics. Medication adherence rates in excess of 100% (e.g., subjects mistakenly took extra pills) will be reported as 100% adherence. Similarly, medication adherence rates below zero (e.g., subjects added pills to the bottle but did not remove any pills) will be reported as 0% adherence. Pill count adherence is an objective measure that has been shown to correlate with electronic monitors and varenicline plasma levels.

CONTACTS AND LOCATIONS:
Overall Officials: Shadi Nahvi, MD, MS, Principal Investigator — Albert Einstein College of Medicine; David Goldfarb, PhD, Principal Investigator — FDNY
Locations (1):
- FDNY World Trade Center Health Program, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data set

REFERENCES:
- [Result] Goldfarb DG, Moline T, Prezant DJ, Bars MP, Zeig-Owens R, Schwartz T, Cannon MF, Vaeth B, Arnsten JH, Webber MP, Nahvi S. Design of a randomized tobacco cessation trial among FDNY World Trade Center responders in a lung cancer screening program. Addict Sci Clin Pract. 2025 Aug 5;20(1):62. doi: 10.1186/s13722-025-00598-3. PMID 40765018